CLINICAL TRIAL: NCT01589016
Title: Single Determination of Serum Activin A and Inhibin A in Predicting the Outcome of Pregnancies of Unknown Location (PUL) After IVF and Oocyte Donation.
Brief Title: Activin A and Inhibin A in Predicting Outcome of Pregnancies of Unknown Location After Assisted Reproductive Technology
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Juan Giles, Gynaecologist IVI Valencia, Instituto Valenciano de Infertilidad, IVI VALENCIA
Other Study IDs: 0711-C-033-JG
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2013-09-19 (Estimated); Status verified 2013-09

CONDITIONS: Ectopic Pregnancies
MeSH Terms: conditions — Pregnancy, Ectopic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — Blood samples are to be taken at the time of the first ultrasound examination and stored at -20ºC. Inhibin A and activin A to be determined by ELISA. β-hCG and P were also determined using Microparticle Enzyme Inmunoassay (MEIA).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- PUL (pregnancy of unknown location),
- EP ( ectopic pregnancies P)
- IUP-singleton intrauterine pregnancies

SUMMARY:
The purpose of this study is to determine the predictive value of a single serum determination of activin A and inhibin A for the prognosis of ectopic pregnancy after in Vitro Fertilization (IVF) cycles, in both native and donated oocytes.

DETAILED DESCRIPTION:
Ectopic pregnancy (EP) is one of the most common pathologies seen in emergency gynaecology practice. Early diagnostic of this situation is a clinical objective because it remains an important cause of maternal morbidity and mortality worldwide. Currently, transvaginal ultrasound scan (TVS) allow ascertain the location of the pregnancy. However, the diagnosis of EP is complicated by a nonspecific clinical presentation and the inconclusive results in some cases of transvaginal ultrasound at first presentation. For this reason several biomarkers have been investigated to accurately detect the establishment of pregnancy and predict its outcome as early as possible.

These biomarkers include: markers of abnormal embryo/trophoblast growth (β-subunit of HCG, Activin A, etc), markers of abnormal corpus luteum function (progesterone, inhibin A, etc), markers of a growing pregnancy in the Fallopian tube (creatine kinase, vascular endothelial growth factor, etc), markers of inflammation and peritoneal irritation (cancer antigen 125, interleukin-6, etc), and uterine markers of normal implantation (leukaemia inhibitory factor and glycodelin). Β-HCG and progesterone are usually used in clinical practice and activin A and inhibin A have recently shown promising results.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pregnancy of unknown location (PUL) diagnosed 22 - 27 days after oocyte retrieval, at first ultrasound routine control (A "pregnancy of unknown location" (PUL) is a term used to classify a women with a positive pregnancy test and an empty uterus with no signs of an intrauterine or extrauterine pregnancy on a transvaginal ultrasound scan.)
* Patients with Intrauterine pregnancy : Viable intrauterine pregnancy (IUP) An intrauterine gestational sac containing a fetal pole with visible cardiac activity
* Patients with Ectopic pregnancy (Tubal ectopic pregnancy): An empty endometrial cavity with: (i) an inhomogeneous adnexal mass or (ii) an empty extrauterine gestational sac seen as hyperechoic ring or (iii) an extrauterine gestational sac with a yolk sac and/or fetal pole with or without cardiac activity

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the first control, made 22-27 days after oocyte retrieval, all women underwent a transvaginal ultrasound (TVS) examination using a 6.5-MHz transducer (Voluson 730 Pro V; General Electric, Madrid, Spain). They were diagnosed with an ectopic pregnancy (EP) or an intrauterine pregnancy (IUP) on the basis of this examination and where there was no clear ultrasound evidence of pregnancy were classified as pregnancy of unknown location (PUL). Women were followed up until the final pregnancy outcome was known.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
levels of activin and inhibin A | within the first two weeks after the first control of pregnancy

SECONDARY OUTCOMES:
Progesterone and BHCG | within the first two weeks after the first control of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Juan Giles, MD, Principal Investigator — IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Valencia, Spain